CLINICAL TRIAL: NCT06054061
Title: Improving Subjective Wellbeing Despite a Severe Psychiatric Condition Through "Think and Cope Positively" Program: A Randomized Control Trial.
Brief Title: Evaluation the Efficacy "Think and Cope Positively" Program
Acronym: PA+
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pontificia Comillas (Other)
Responsible Party: Principal Investigator, Rocio Caballero Campillo, Assistant Collaborator - Clinical Professor, Universidad Pontificia Comillas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7/22-23; CX22-00110 (Other Grant/Funding Number: Fundación "la Caixa")
Record Dates: First submitted 2023-09-05; First posted 2023-09-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Mental Disorder
Keywords: Schizophrenia; Subjective Well-Being; Optimism; Coping; Purpose of life
MeSH Terms: conditions — Mental Disorders; Schizophrenia

STUDY DESIGN:
Intervention Model Description: A multicenter cluster randomized clinical trial will be conducted. The trial will consist of two arms, the experimental group will receive a 15-week intervention based on the promotion of hedonic and eudaimonic well-being. The control group will remain on a waitlist with their Treatment as Usual. Participants will be recruited from centers that focus on the psychosocial rehabilitation of people diagnosed with schizophrenia spectrum, bipolar disorder, personality disorders and severe affective disorders. Random allocation to the groups will be stratified according to the typology of the center. In the event that there is only a single representative of one of the center typologies, the entire center will be assigned to one of the study conditions. Assessments will be made before the intervention (E1), immediately after the 15-week intervention period (E2) and three (E3) and six (E4) months after the end of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAU + Wellbeing promotion group (Think and Cope Positively) Intervention (Experimental): In addition to their usual treatment, participants form the experimental arm will receive 15 weekly intervention sessions, where aspects related to subjective wellbeing, life plans, alliance with the therapist or family and social relationships will be worked on.
  Interventions: Behavioral: Experimental: experimental wellbeing promotion group (Think and Cope Positively); Behavioral: TAU
- TAU + waiting list (Other): The control group will continue to receive the treatment as usual in their intervention resources. At the end of the 15-week control period they will receive the intervention.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Experimental: experimental wellbeing promotion group (Think and Cope Positively) — Session 1: Welcome. 2: Identifying and amplifying positive emotions. 3: Experiencing positive emotions. 4: Identifying my negative "trap" thoughts. 5: Transforming my automatic thoughts into positive ones. Session 6: Experiencing my positive thoughts I. 7: Experiencing my positive thoughts II. 8: Learning to be kinder to myself. 9: Identifying a life project (Individual appointment).10: Identifying coping strategies I. 11: Identifying coping strategies II. 12: Identifying adaptive coping strategies linked to well-being. 13: Building my life purpose with my environment. 14: Helping me to build my life purpose? 15: Multi-family session, farewell and closing.
  Arms: TAU + Wellbeing promotion group (Think and Cope Positively) Intervention
Behavioral: TAU — The usual treatment in the intervention of people affected by severe mental disorder in the network of public and subsidized centers in Spain consists of improving psychosocial functioning. To this end, and depending on the characteristics of the user, work is done in groups and individually on social skills, psychoeducation about the disease, adherence to pharmacological treatment, improvement of daily living activities, promotion of independent leisure, support to families in the process of relapse prevention, and training for labor market insertion.

SUMMARY:
The purpose of this study is to determine whether an integrated protocol based on cognitive behavioural therapy, positive psychology and third generation therapies is effective in improve the subjective well-being of people affected by a severe mental illness (SMI).

The design of the study is a cluster randomized control trial with two arms. Experimental groups will receive 15 sessions to enhance positive emotions, optimism, adaptive coping, finding a purpose in life and sharing it with people who are important to the user. The control group will remain on a waitlist with their treatment as usual (TAU). After the control period (15 weeks), participants of the experimental groups have the chance to receive the intervention. Both groups will be measure before and after de 15 intervention weeks. Additionally, follow-up measures of the experimental group will be taken after 3 and 6 months.

DETAILED DESCRIPTION:
This research aims to generate evidence on the usefulness of interventions focused on the well-being of people diagnosed with SMI, trying to alleviate some of the limitations found in previous protocols.

Regarding the content of the sessions, optimism, low levels of depression, social support and the degree of agreement with the therapist, have recently been identified as the factors that best predict subjective well-being in people affected by SMI. Therefore, modules on optimism and coping focused on well-being will be included, maintaining the emphasis of the work on positive emotions. By adding an individual work session in which goals and objectives are agreed upon by the therapist and user, the consensus will be strengthened between both parties. After discussing the construction of a life project throughout the protocol, the process the process will conclude with a session combined users and the special persons chosen by the participants. Both members will have the opportunity to share with each other.

Finally, we will follow the indications of recent studies which demonstrate that, in order to improve the optimistic response in psychiatric populations, it is necessary to reformulate negative thinking, practice hopeful thinking, practice gratitude and build a life project.

ELIGIBILITY:
Inclusion Criteria:

* Users of public psychosocial rehabilitation resources belonging to the Community of Madrid and Castilla la Mancha
* Legal age
* Clinical diagnosis of severe mental disorder: schizophrenia spectrum, bipolar disorder, personality disorders and severe affective disorders.
* Psychopathological stability (or that residual symptoms do not interfere with the course of treatment)
* Minimum level of cognitive comprehension (i.e. no comorbidity with intellectual disability).

Exclusion Criteria:

* Addiction dependence criteria (on the other hand, people with substance abuse criteria will be accepted)
* Altered behavior (relationally) that could alter the good functioning of the group.

Prior to their participation in the study, the rehabilitation team, in coordination with the research team, will assess whether the patient can benefit from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with life scale (SWLS) | This test is applied before starting the intervention protocol, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  The scale evaluate hedonic well-being by 5 items with a 7-point Likert-type response scale (strongly disagree - strongly agree). Mean scores range from 1 to 5. Higher scores indicates higher hedonic well being.
Psychological Well-being Scale (SPWB) | This test is applied before starting the intervention protocol, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  The scale evaluate eudaemonic well-being by 29 items with a Likert-type scale from 1 to 6 (totally disagree - totally agree). The scale measures 6 domains of well being (self-acceptance, purpose in life, personal growth, positive relationships, autonomy and mastery of the environment). Mean scores range from 1 to 6. Higher scores indicates higher eudaemonic well being or domain.

SECONDARY OUTCOMES:
Openness to the Future Scale (OFS) | This test is applied before starting the intervention protocol, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  This scale evaluate optimism conceptualized as a positive affective state by 10 items with a Likert-type scale from 1 to 6 (totally disagree - totally agree). Mean scores range from 1 to 6. Higher scores indicates higher optimism.
Therapeutic Alliance and Theory of Change Inventory (WATOCI) | This test is applied before starting the intervention protocol, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  This scale evaluate the alliance with the therapist by 17 items with a Likert-type scale from 1 to 7 (never - always). Mean scores range from 1 to 7. Higher score indicates higher alliance with the therapist.
Symptom Checklist-45 abbreviated version | This test is applied before starting the intervention protocol, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  This test evaluates psychological symptom by 45-items with a Likert-type scale from 0 to 4 (Not at all - Very much or extremely). The scale evaluates 9 domains (Depression, Hostility, Interpersonal sensitivity, Somatization, Anxiety, Psychoticism, Obsession-Compulsion, Phobic anxiety and, Paranoid ideation). Mean scores range from 0 to 4. A higher score indicates more intense symptoms.

OTHER OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | This test is applied before starting the intervention protocol, at the end of each of the 15 intervention sessions, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  This scale enable the monitoring of mental wellbeing in the general population and is frequently used in evaluation of projects, programs and policies which aim to improve mental wellbeing. The scale presented seven items, answered in a 5-point Likert scale from 1 to 5 (never - always or almost always). Mean scores range from 1 to 5. Higher scores indicates higher wellbeing.
Clinical Outcomes in Routine Evaluation-Outcome Measure-5 (CORE-OM) | This test is applied before starting the intervention protocol, at the end of each of the 15 intervention sessions, immediately after the end of the 15-week intervention protocol, and at 3 and 6 months after the end of the intervention protocol.
  The brief form of the CORE-OM assesses psychological distress by 5 items, which present a 5-points Likert-type scale from 0 to 4 (never - always or almost always). Mean scores range from 0 to 4. Higher scores indicates higher psychological distress.
Protocol adherence form | This record is applied by the therapist at the end of each of the 15 intervention sessions. This measure will be carried out after each treatment session assessed up to 24 months
  At the end of each session, the group therapists fill out a 10-item inventory in which they indicate the fulfillment of the session's objectives using a 3-points Likert scale 0 to 2 (not achieved - partially achieved - fully achieved).
Attendance and exercise engagement form | This record is applied by the therapist at the end of each of the 15 intervention sessions. This measure will be carried out after each treatment session assessed up to 24 months
  At the end of each session, the therapists record the participants who attended the session and the performance of the exercises at home before the session and in the session.
Participants' satisfaction was measured by the Client Satisfaction Questionnaire (CSQ-8, Larsen et al., 1979). | This register is applied at the end of the 15-week intervention period.
  The CSQ-8 is an 8-item measure that assessed general satisfaction with the group by a 4-points Likert-type scale from 1 to 4 (very dissatisfied - very satisfied). Mean scores range from 1 to 4. Higher scores indicate higher satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Caballero-Campillo, Dra, Principal Investigator — UNINPSI, Universidad Pontificia Comillas
Locations (1):
- UNINPSI, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No